CLINICAL TRIAL: NCT02423421
Title: Randomised Placebo Controlled Trial of Faecal Microbiota Transplantation in Irritable Bowel Syndrome
Brief Title: Faecal Microbiota Transplantation in Irritable Bowel Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Professor Fergus Shanahan, Professor and Chair Department of Medicine and Director Alimentary Pharmabiotic Centre, University College Cork, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APC053
Record Dates: First submitted 2015-03-10; First posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Active Comparator): The treatment group will have faecal microbiota transplantation performed using stool from a healthy human donor
  Interventions: Other: Faecal microbiota transplantation
- Placebo group (Placebo Comparator): The placebo group will have autologous faecal microbiota transplantation performed.
  Interventions: Other: Faecal microbiota transplantation

INTERVENTIONS:
Other: Faecal microbiota transplantation — Human Stool.

SUMMARY:
The purpose of thus study is to determine if faecal microbiota transplantation will result in improvement in clinical outcomes in patients with irritable bowel syndrome.

DETAILED DESCRIPTION:
1. Background

   Irritable bowel syndrome (IBS) is a chronic, debilitating, functional gastrointestinal disorder with estimated population prevalence in Europe between of 10 -15% (Ford et al). These symptoms can be debilitating and lead to a significant reduction in quality of life particularly in the more severely affected.

   Alterations in the function and composition of the gut microbiota are increasingly being implicated as potential aetiological factors. (Collins et al). One of the strongest indictors for this concept is the significantly increased risk of developing IBS after an episode of acute gastroenteritis. Prospective studies have demonstrated that between 3- 36% of enteric infections lead to new, persistent IBS symptoms. (Gwee at al.,Neal et al) A number of studies have demonstrated that the diversity, stability and metabolic activity of the gut microbiota are altered in IBS patients compared with healthy individuals (Jeffrey et al). Although a distinct microbial signature has not been identified for IBS, several studies have shown a gut microbial composition enriched with Firmicutes together with a reduced abundance of Bacteroides (Jeffery et al, Rajilic-Stojanovic et al).

   Faecal microbial transplantation (FMT) has proven to a safe, inexpensive and effective treatment for recurrent Clostridium difficile infection achieving up to 90% cure rates in some studies with a very good side effect and adverse event profile (van. Nood et al.). In this study the investigators wish to investigate whether restoring healthy gut microbiota profiles, using stool from healthy donors, will lead to improved clinical outcomes for patients with IBS.

   Autologous fecal microbiota transplant using re - infusion of the participants own faeces has been previously been used as a placebo in studies using FMT (Vrieze et al)
2. Study Design

   The design of the study is a prospective randomised, placebo controlled study that will be carried out on a single site. The study will involve four visits in total over an 8 week period. The first visit will be a screening visit to assess eligibility for the study. Visit two will be the treatment visit at which patients will receive the FMT using stool from a healthy donor or placebo. An autologous faecal microbiota transplant will be used as the placebo in this study. Follow up visits will be performed at 4 weeks and 8 weeks after the treatment.

   Up to 50 patients with IBS will be recruited for the study. All patients will have an established diagnosis of IBS as per the Rome III criteria. Subjects will be recruited from the population of IBS patients attending Cork gastroenterology outpatients. Subjects will be randomly assigned to either the treatment group or placebo control group.
3. Donor Selection:

   Donor stool will be obtained from healthy donors. The donors will be interviewed to ensure they are in good health and will undergo a screening questionnaire to identify potential infectious risk which could be transferred by stool. Certain exclusion criteria will apply and donors will undergo testing of stool and serum. The donation process is safe for the donor (Bakken et al). A selected healthy individual with a diverse microbial composition will preferentially be used as the donor candidate unless recipient wishes dictate the use of a designated donor.

   3.1 Donor Exclusion criteria

   Risk of infectious agent Known Human immunodeficiency virus, hepatitis B or C. Known exposure to HIV or viral hepatitis Known current communicable disease High risk lifestyle factors Factors which increase risk of Creutzfeldt-Jakob disease. Gastrointestinal co-morbidities History of inflammatory bowel disease History of IBS History of gastrointestinal malignancy or polyposis History of major Gastrointestinal surgery Factors that can or do affect the composition of the intestinal microbiota. Antibiotics within the preceding 3 months Major immunosuppressive medications Systemic anti-neoplastic drugs Additional recipient specific considerations Recent ingestion of a potential allergen where recipient has a known allergy. Systemic autoimmunity Atopic diseases Chronic pain syndrome Obesity.

   3.2 Donor Testing

   The following screening tests will be performed on all potential donors:

   Stool testing Clostridium difficile by polymerase chain reaction (PCR) PCR for Shigella, Salmonella, E.coli verotoxin, Campylobacter Cryptosporidium Ova and parasites Serological testing HIV, type 1 and 2 Hepatitis A IgM Hepatitis B surface antigen, hepatitis B core antibody and hepatitis B surface antibody.

   Hepatitis C screen human T-cell leukemia virus (HTLV) Rapid Plasma Reagin and fluorescent treponemal antibody absorbed.
4. FMT procedure protocol:

The following procedures should be followed in terms of donor and recipient preparation and in the preparation and administration of the donor stool.

1. Donor Preparation Can use gentle osmotic laxative the night before procedure. Provide the stool sample on the morning of the procedure.
2. Recipient Preparation Standard pre colonoscopy bowel preparation on the day before the FMT.
3. Stool preparation After passage of the stool by the donor it will be immediately be transferred to an anaerobic hood to be processed.

   The stool will be diluted and filtered producing a liquid slurry consistency The liquid stool will then be placed in an anaerobic bottle and transferred to the site of administration.
4. Stool administration. The stool should be administered as soon as possible after it's prepared, at maximum 2 hours.

   The FMT will be performed endoscopically. All patients will undergo a colonoscopy and the liquid stool will be infused through the endoscope.

   Ideally all patients will also have a duodenal infusion of stool performed via an oesphogastrodoudenoscopy at the same session. However if the patient does not consent to this it will not be deemed a protocol breach.
5. Study Procedures:

   The study will be conducted as outlined in this protocol and in accordance with the ICH Guidelines on Good Clinical Practice, and the declaration of Helsinki [Appendix A]. Informed consent will be obtained prior to any study related procedures being undertaken.

   5.1.1 Screening Visit (Visit 1)

   The aim of the study and the procedures to be undertaken will be explained to all potential subjects. Subjects will then be requested to read the subject information sheet and read and sign the informed consent form, and will receive a signed copy. The following assessments will be performed at Visit 1 Informed consent Demographics Medical and medication history Rome III questionnaire Evaluation of eligibility criteria Vital signs Physical examination, body weight, height and BMI assessment Food frequency questionnaire IBS symptom assessment scores Hospital Anxiety and Depression Scale International Physical activity Index Blood samples Stool samples

   If the patient meets the eligibility criteria they will return within 28 days to undergo faecal microbiota transplantation.

   5.1.2 Treatment Visit (Visit 2)

   At visit 2 the patients will undergo faecal microbial transplantation. Prior to the procedure all patients should undergo standard bowel preparation. At Visit 2 the following assessments will be performed on all patient before FMT is performed Brief interview about the previous weeks Vital signs and physical examination. Eligibility assessment Informed consent for endoscopy.

   The donor stool will be administered to the patient endoscopically. All patients will undergo colonoscopy and the donor stool will be infused through the colonoscope. Decision to perform duodenal infusion as well as colonic infusion will be dictated by patient preference. If the patient consents they will also undergo oesphogastrodoudenoscopy and donor stool will be infused through the gastroscope into the patients duodenum.

   Following the procedure the patent will be managed in recovery as per standard endoscopy guidelines.

   5.1.3 Visit 3 and 4 - Follow up visits.

   At visits 3 and 4 the patients will undergo the following Interview about the previous weeks. Vital signs and physical exam incl BMI Concomitant medication Adverse events monitoring Blood samples for clinical and research. Stool sample (collected at home prior to visit). Food frequency questionnaire IBS symptom assessment scores Global assessment question. Hospital Anxiety and Depression Scale International Physical activity Index

   5.2 Removal of subjects from the study

   Subjects will be withdrawn from the study if the subject; Elects independently to withdraw from the study; If he/she develops any condition which contravenes the original criteria; Is considered at any point to be unsuitable to continue the study, at the discretion of the investigator.

   5.3 Concomitant Medication

   Subjects will be questioned about their medication history. The details of any medication taken will be recorded in the patient case notes and case report form

   5.4 Endpoint assessments

   Subjects will have the following endpoint assessments performed: assessment of medical and surgical history changes since baseline/treatment visits, IBS severity/QOL scores, faecal sample assessment/analysis, blood sample analysis, physical assessment, concomitant medication and adverse events.

   To ensure subject safety the following evaluations will be performed during the study: vital signs, adverse event monitoring, physical examination and laboratory assessments
6. Biological Sample Collections and Analysis:

6.1 Blood

Blood will be collected at each visit for clinical haematological and biochemical analysis and cytokine analysis.

Haematology and biochemistry panels will be done as per standard of a care - Full blood counts (including haemoglobin, white cell count, platelet count, haematocrit and differential white cell count), erythrocyte sedimentation rate(ESR), sodium, potassium, chloride, urea, creatinine, protein, albumin, crp, liver function tests and quantitative immunoglobulin (IgA, Immunoglobulin G, IgM). Participants will also have HIV, hepatitis B, hepatitis C, HTLV and syphilis screens performed at visit 1. This analysis will be performed at Cork University Hospital (CUH) laboratories. All laboratory results will be reviewed and reports signed the investigators and recorded in the patients case repot form (CRF).

Research bloods for serum analysis of inflammatory immune markers including cytokines will be performed, theses bloods will be processed in the laboratories of the Alimentary Pharmabiotic Centre, University College Cork(UCC).

6.2 Faecal Sample

Faecal samples will be collected at each visit. Bacterial DNA will be extracted from the faecal samples of each subject and the composition of the microbiota determined by sequencing of amplified bacterial ribosomal ribonucleic acid (RNA) genes, before and after the faecal microbiota transplantation is performed. Faecal samples will also be analysed for viral particles and phageome studies performed.

6.3 Biopsy/ Intestinal Tissue Collections, Storage and Analysis

If the patient consents, during their endoscopy at time of FMT biopsy of intestinal tissue will be performed. The tissue samples will be collected in culture medium and stored at 4 0C until delivered to the lab in UCC. Microbiota composition analysis will be performed by direct pyrosequencing of 20,000-40,000 16S rRNA gene amplicons per subject (Pubmed: 20571116). Sequence generation and analysis performed by the UCC bioinformatics team will determine the composition of the microbiota of individuals.

6.4 Analyses

Analyses of all samples collected will be conducted in the CUH and/or UCC/Teagasc laboratories. On some occasions the analyses may be done in collaboration with a third party outside UCC including pharmaceutical companies, which may require samples to be shipped to this organisation. These samples will be coded and identified only using anonymised sample identifier numbers. In addition samples may be stored and used for analysis in future studies. Again samples will be coded and identified only using anonymized sample identifier numbers.

7 .Statistics and Study Powering:

A placebo response rate of 40% is predicted in this study population. The study will be appropriately powered to detect additional benefit of at least 15% in the treatment group compared to placebo.

The primary and secondary objectives will be analysed using standard parametric and non-parametric statistical techniques to test the efficacy of FMT. The exploratory objective will be assessed using sophisticated biostatistical analysis to identify a microbiota profile that predicts response to FMT.

8. Changes in the conduct of the study or planned analyses:

With the exception of emergency situations, any significant change in the protocol (i.e., one that affects the safety of the subjects, scope of the investigation, the scientific quality of the study) will not be implemented until the Independent Ethics Committee (IEC) have reviewed, approved, and documented the protocol amendment in writing. Amendments include changes in the investigator and investigators or site address, etc.

When a change is made to eliminate or reduce the risk to subjects, it may be implemented before review and approval by the IEC. The investigator shall notify the IEC of said change in writing within 5 working days after implementation.

In the event of an emergency, the investigator shall institute any medical procedures deemed appropriate, however all such procedures (minor or non significant), change (e.g. Statistician, typographical errors, spelling errors, etc) will not be made until said change is reviewed and approved by the Independent Ethics Committee and a memo communicating the change is provided by the investigator.

9. Obligation of the investigator:

The study will be conducted in accordance with the applicable Good Clinical Practice 21 Code of Federal Regulations 50, 56, and 312; International Conference of Harmonisation (ICH) Good clinical practice published in the Federal register; 9 May 97 (volume 62,number 90, pages 25691-25709).

The investigator will perform or directly supervise the performance of all the services described herein, or incidental to those described herein, in accordance to the highest standards of medical and clinical research practice. Delegation of any study responsibility will be documented in writing.

It is the responsibility of the investigator and any co-investigator to understand and follow the protocol, and to ensure that all the members of the assisting staff also understand and follow the protocol.

10. Advertising:

All advertisements for subjects, whether in a professional or consumer publications, radio, television, or any other means, will be approved by the Independent Ethics Committee prior to initiation.

11. Institutional review:

The site, investigator, protocol, informed consent form and any other pertinent documents for this study will be approved by:

Cork Research Ethics Committee of the Cork Teaching Hospitals, Lancaster Hall, 6 Little Hanover Street, Cork.

The study will not begin until the IEC has approved of the protocol and the subject consent form along with any advertisements, diaries and instructions to the subjects, if applicable. The IEC approval will be documented in writing to the investigator.

12. Subject Consent:

Independent Ethics Committee approval of the written informed consent will be obtained prior to its use.

This consent form will comply with all the regulations governing the protection of human subjects.

Each subject will sign and date an informed consent form to serve as a participant in the study. A signed copy of the consent form will be given to the subject and a signed copy will be retained by the investigator in the patient's case notes.

Subjects may withdraw from participation in the study at any time without detriment. Additionally, the investigator may withdraw subjects from the study if it is in the best interest of the subjects. The reason for subject withdrawals from the study will be documented in the subject's case notes.

13. Data Collection:

All data collected will be entered in the subjects case report form and computer database, it will be handled and stored safely in confidential conditions. Study records will be stored in a locked metal filing cabinet in a locked office in Cork University Hospital and in computer databases, which require entry code.

The investigator has the responsibility for ensuring that all source documents (i.e. study and/ or medical records) are completed and maintained according to the study protocol and Good Clinical practice and is available at the site.

Source documents for this study will include hospital records and procedure reports and data collection forms. These documents will be used to enter data on the CRFs.

All conventional precautions will be maintained to ensure documents will be stored safely in confidential conditions. The identity of all patients' samples and study records other than the signed consent will be coded and computer databases will adopt codes rather than patient names. In addition, computer access will require entry code.

If for any reason, the subject does not complete the study, an explanation will be entered on the case notes.

Data entry/management methods will be in accordance with the study protocol and Good Clinical Practice. The identity of all study subjects will be by individual study numbers. The name or any other identifying details of the subjects will not be included in any study data electronic file or CRF

14. Institutional review:

The site, investigator, protocol, informed consent form and any other pertinent documents for this study will be approved by:

Cork Research Ethics Committee of the Cork Teaching Hospitals, Lancaster Hall, 6 Little Hanover Street, Cork.

The study will not begin until the IEC has approved of the protocol and the subject consent form along with any advertisements, diaries and instructions to the subjects, if applicable. The IEC approval will be documented in writing to the investigator.

15. Finance and Insurance policy:

This study is being sponsored by the Alimentary Pharmabiotic Centre, University College Cork, and will be indemnified by University College Cork's liability coverage for human research.

16. Adverse and Serious adverse events:

Adverse events and serious adverse events will be monitored and recorded throughout the study to ensure patient safety.

At each visit, subjects will be queried about any adverse events they may have experienced since the last visit.

All adverse events (AEs) reported will be coded using the COSTART5 dictionary and listed documenting duration, severity, relationship to study treatment, subject outcome, and if any therapy was required.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrolment into the study, subjects must;

* Be able to give written informed consent.
* Males and females aged >18 and <65
* Have IBS as defined by the Rome III criteria

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the below criteria;

* Are less than 18 and greater than 65 years of age.
* Have a significant acute or chronic coexisting illness (cardiovascular, gastrointestinal, endocrine, immunological, metabolic or any condition which contraindicates, in the investigators' judgment, entry to the study).

Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.

* Are receiving treatment involving experimental drugs.
* If the subject has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study.
* Have a malignant disease or any concomitant end-stage organ disease Pregnancy
* Use of antibiotics within 6 weeks of screening.
* Use of systemic steroids within the last month.
* Use of an antipsychotic within prior 3 months.
* Have suffered from a major psychiatric disorder with the past two years.
* Lactose intolerance.
* Those > 55 will be excluded if they have not had a sigmoidoscopy or colonoscopy within previous 5 years.
* Any abdominal surgery other than hernia repair or appendicectomy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Global Assessment of relief of IBS symptoms. | 8 weeks
  This assessment will be obtained by defining the response (Yes or No) to the following question.
  "Please consider how you felt in the past week in regard to your IBS, in particular your overall well-being, and symptoms of abdominal discomfort or pain, bloating or distension and altered bowel habit .Compared to the way you usually felt before the beginning of the trial, have you had adequate relief of your IBS-symptoms?"

SECONDARY OUTCOMES:
Primary symptoms of IBS | 8 weeks
  The primary symptoms of IBS will be scored on a six point Likert scale at baseline, week 4 and at end of study. The following symptoms will be assessed and recorded: abdominal pain/discomfort, bloating/distension, sense of incomplete evacuation, straining at stool, urgency of bowel movement, passage of gas and mucus, bowel habit satisfaction. Each symptom will be assessed using a 6-point scale, where 0 = none to 5 = very severe. Bowel habit satisfaction will be assessed using a 6-point scale where 0 = very satisfied and 5 = very dissatisfied. Overall assessment of IBS symptoms will be also be scored on a 6 - point scale. An IBS composite score(15 point score) representing the sum of individual scores for abdominal pain/discomfort, bloating/distension, and bowel movement difficulty (straining at stool or urgency of bowel movement) will be calculated.
Quality of life | 8 weeks
  At baseline and at the end of the study each subject will complete an IBS-specific quality of life questionnaire (IBS-QOL)
Depression and Anxiety | 8 weeks
  At baseline and at the end of the study each subject will complete the Hospital Anxiety and Depression (HAD) Scale.
Safety as measured by occurrence of adverse events | 8 weeks
  Patients will be monitored throughout the study period and they will be recorded as per the The Consolidated Standards of Reporting Trials (CONSORT) criteria

OTHER OUTCOMES:
Patient microbiota compositional profiles | 8 weeks
  We will characterise all participants' microbiota composition at baseline and at the end of study to determine if there is a subgroup of patient/donor combinations, based on their microbiota composition, in whom a positive response to FMT was obtained. This would be very valuable for future optimization of a positive primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Fergus Shanahan, MD, DSc, Principal Investigator — Professor and Chair Dept. of Medicine, University College Cork
Locations (1):
- Alimentary Pharmabiotic Centre, University College Cork, Cork, Cork, Ireland

REFERENCES:
- [Background] Drossman DA, Camilleri M, Mayer EA, Whitehead WE. AGA technical review on irritable bowel syndrome. Gastroenterology. 2002 Dec;123(6):2108-31. doi: 10.1053/gast.2002.37095. No abstract available. PMID 12454866
- [Background] Gwee KA, Graham JC, McKendrick MW, Collins SM, Marshall JS, Walters SJ, Read NW. Psychometric scores and persistence of irritable bowel after infectious diarrhoea. Lancet. 1996 Jan 20;347(8995):150-3. doi: 10.1016/s0140-6736(96)90341-4. PMID 8544549
- [Background] Collins SM. A role for the gut microbiota in IBS. Nat Rev Gastroenterol Hepatol. 2014 Aug;11(8):497-505. doi: 10.1038/nrgastro.2014.40. Epub 2014 Apr 22. PMID 24751910
- [Background] Ford AC, Talley NJ. Irritable bowel syndrome. BMJ. 2012 Sep 4;345:e5836. doi: 10.1136/bmj.e5836. No abstract available. PMID 22951548
- [Background] Neal KR, Barker L, Spiller RC. Prognosis in post-infective irritable bowel syndrome: a six year follow up study. Gut. 2002 Sep;51(3):410-3. doi: 10.1136/gut.51.3.410. PMID 12171965
- [Background] Jeffery IB, Quigley EM, Ohman L, Simren M, O'Toole PW. The microbiota link to irritable bowel syndrome: an emerging story. Gut Microbes. 2012 Nov-Dec;3(6):572-6. doi: 10.4161/gmic.21772. Epub 2012 Aug 16. PMID 22895081
- [Background] Rajilic-Stojanovic M, Biagi E, Heilig HG, Kajander K, Kekkonen RA, Tims S, de Vos WM. Global and deep molecular analysis of microbiota signatures in fecal samples from patients with irritable bowel syndrome. Gastroenterology. 2011 Nov;141(5):1792-801. doi: 10.1053/j.gastro.2011.07.043. Epub 2011 Aug 5. PMID 21820992
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Kassam Z, Lee CH, Yuan Y, Hunt RH. Fecal microbiota transplantation for Clostridium difficile infection: systematic review and meta-analysis. Am J Gastroenterol. 2013 Apr;108(4):500-8. doi: 10.1038/ajg.2013.59. Epub 2013 Mar 19. PMID 23511459
- [Background] Gough E, Shaikh H, Manges AR. Systematic review of intestinal microbiota transplantation (fecal bacteriotherapy) for recurrent Clostridium difficile infection. Clin Infect Dis. 2011 Nov;53(10):994-1002. doi: 10.1093/cid/cir632. PMID 22002980
- [Background] Bakken JS, Borody T, Brandt LJ, Brill JV, Demarco DC, Franzos MA, Kelly C, Khoruts A, Louie T, Martinelli LP, Moore TA, Russell G, Surawicz C; Fecal Microbiota Transplantation Workgroup. Treating Clostridium difficile infection with fecal microbiota transplantation. Clin Gastroenterol Hepatol. 2011 Dec;9(12):1044-9. doi: 10.1016/j.cgh.2011.08.014. Epub 2011 Aug 24. PMID 21871249
- [Background] Vrieze A, Van Nood E, Holleman F, Salojarvi J, Kootte RS, Bartelsman JF, Dallinga-Thie GM, Ackermans MT, Serlie MJ, Oozeer R, Derrien M, Druesne A, Van Hylckama Vlieg JE, Bloks VW, Groen AK, Heilig HG, Zoetendal EG, Stroes ES, de Vos WM, Hoekstra JB, Nieuwdorp M. Transfer of intestinal microbiota from lean donors increases insulin sensitivity in individuals with metabolic syndrome. Gastroenterology. 2012 Oct;143(4):913-6.e7. doi: 10.1053/j.gastro.2012.06.031. Epub 2012 Jun 20. PMID 22728514